CLINICAL TRIAL: NCT01700829
Title: Ketamine vs. Midazolam: Testing Rapid Relief of Suicide Risk in Depression
Brief Title: Ketamine in the Treatment of Suicidal Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Grunebaum, MD, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #6598; R01MH096784 (NIH)
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Major Depressive Disorder; Suicidal Ideation
Keywords: Ketamine; Midazolam; Major Depressive Disorder; Suicidal ideation; Suicide; Depression; Treatment; Ketamine Treatment
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation; Suicide; Depression | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midazolam (Active Comparator): 0.02 mg/kg, I.V. (in the vein)
  Interventions: Drug: Midazolam
- Ketamine (Active Comparator): 0.5 mg/kg, I.V. (in the vein)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Single dose of 0.5 mg/kg of ketamine given intravenously (in the vein) over 40 minutes
  Other Names: Ketalar; Ketamine Hydrochloride Injection
  Arms: Ketamine
Drug: Midazolam — Single dose of 0.02 mg/kg of Midazolam given intravenously (in the vein) over 40 minutes
  Other Names: Midazolam Injection
  Arms: Midazolam

SUMMARY:
This study is designed to compare the effectiveness of two medications, Ketamine and Midazolam, for rapidly relieving suicidal thoughts in people suffering from depression.

The first drug, Ketamine, is an experimental antidepressant that early studies have shown may quickly reduce suicidal thoughts, but we are not sure how well it may work. Midazolam, the comparison drug, is not thought to reduce depression or suicidal thoughts.

DETAILED DESCRIPTION:
Patients currently taking psychiatric medications may continue them during the study. However, if a patient is taking a benzodiazepine (such as Ativan, Klonopin, or Xanax), they will be able to take up to 2mg per day of Lorazepam during the week before the infusion, but none will be permitted in the 24 hours pre-infusion. Also, Zolpidem (Ambien) will not be permitted in the 24 hours pre-infusion. If a person chooses to participate, their dose of benzodiazepine may need to be reduced so that they can do without it during the 24 hours pre-infusion.

Depressed participants are randomly assigned to receive a single dose of Ketamine(0.5 mg/kg) or Midazolam (0.02 mg/kg), which is given slowly, in a vein, over about 40 minutes. The study is "double-blind," meaning patients and study staff will not know which medication is in the infusion.

If a patient does not respond to the first infusion, and s/he received Midazolam, then s/he will be offered the option of a second infusion, this time with Ketamine (0.5 mg/kg). S/he will then start treatment with a standard antidepressant, unless s/he is not already taking one.

After the infusion(s), participants will have weekly research interviews for 6 weeks to monitor response.

If a patient does have a sufficient infusion response, and s/he is not already taking an antidepressant, then s/he will receive 6-weeks antidepressant research treatment with Sertraline, Fluoxetine, Paroxetine, or Escitalopram, followed by open clinical treatment. However, if s/he is already taking an antidepressant, then s/he will receive open treatment. If s/he does not have a sufficient infusion response, then s/he will receive open treatment.

Participation in this study requires a brief inpatient stay, at no cost, at the New York State Psychiatric Institute (NYSPI).

Eligible participants enrolled in this study will be offered medication management visits at no cost for a total of up to 6 months from the date of enrollment combining inpatient and outpatient treatment. Study medications (Sertraline, Fluoxetine, Paroxetine, Escitalopram, Lorazepam, Zolpidem) will be at no cost during the 6 months. The study will not provide other medications at no cost.

ELIGIBILITY:
INCLUSION CRITERIA:

* Unipolar depression with current major depressive episode (MDE). Participants may be psychiatric medication-free, or if on psychiatric medication, not responding adequately given current MDE with suicidal ideation (See 2).
* Moderate to severe suicidal ideation
* 18-65 years old
* Participants must agree to a voluntary admission to an inpatient research unit at the New York State Psychiatric Institute (NYSPI)for the infusion(s), for a brief stay, or longer if clinically necessary.
* Pre-menopausal female participants of child-bearing potential must be willing to use an acceptable form of birth control during study participation such as condoms, diaphragm, or oral contraceptive pills.
* Able to provide informed consent
* Participants 61-65 years old must score a 25 or higher on the Mini-Mental State Examination (MMSE) at screening.

EXCLUSION CRITERIA:

* Unstable medical condition or neurological illness, including baseline hypertension (BP>140/90) or significant history of cardiovascular illness.
* Significant ECG abnormality
* Pregnant or lactating
* Diagnosis of bipolar disorder or psychotic disorder
* Contraindication to any study treatment.
* Inadequate understanding of English.
* Prior ineffective trial of or adverse reaction to Ketamine or Midazolam.
* Opiate use greater than total daily dose of 20mg Oxycodone or equivalent during the 3 days pre-infusion.
* A diagnosis of sleep apnea.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-06; Primary Completion 2017-01-12 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Grunebaum, M.D., Principal Investigator — Columbia University/New York State Psychiatric Institute
Locations (1):
- Columbia University/New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Hochschild A, Keilp JG, Madden SP, Burke AK, Mann JJ, Grunebaum MF. Ketamine vs midazolam: Mood improvement reduces suicidal ideation in depression. J Affect Disord. 2022 Mar 1;300:10-16. doi: 10.1016/j.jad.2021.12.055. Epub 2021 Dec 22. PMID 34953926
- [Derived] Keilp JG, Madden SP, Marver JE, Frawley A, Burke AK, Herzallah MM, Gluck M, Mann JJ, Grunebaum MF. Effects of Ketamine Versus Midazolam on Neurocognition at 24 Hours in Depressed Patients With Suicidal Ideation. J Clin Psychiatry. 2021 Nov 2;82(6):21m13921. doi: 10.4088/JCP.21m13921. PMID 34727422
- [Derived] Grunebaum MF, Mann JJ, Galfalvy HC, Gibbons RD. Computerized-Adaptive vs. Traditional Ratings of Depression and Suicidal Thoughts: An Assay Sensitivity Pilot Study in a Ketamine Clinical Trial. Front Psychiatry. 2021 Apr 7;12:602976. doi: 10.3389/fpsyt.2021.602976. eCollection 2021. PMID 33897480
- [Derived] Grunebaum MF, Galfalvy HC, Choo TH, Keilp JG, Moitra VK, Parris MS, Marver JE, Burke AK, Milak MS, Sublette ME, Oquendo MA, Mann JJ. Ketamine for Rapid Reduction of Suicidal Thoughts in Major Depression: A Midazolam-Controlled Randomized Clinical Trial. Am J Psychiatry. 2018 Apr 1;175(4):327-335. doi: 10.1176/appi.ajp.2017.17060647. Epub 2017 Dec 5. PMID 29202655
- See also: Additional Information — https://sites.google.com/site/ketamineinsuicidaldepression/
- See also: MIND Clinic for Mood and Personality Disorders — http://www.columbiapsychiatry.org/mind/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Midazolam | Ketamine
Started | 41 | 41
Completed | 40 | 40
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Ketamine | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (13.1) | 38.4 (13.2) | 39.5 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 14 | 18 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 39 | 40 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 39 | 35 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Scale for Suicidal Ideation [Mean (Standard Deviation); unit: units on a scale] — The clinician-rated version of the Beck Scale for Suicidal Ideation was used to assess current severity of suicidal ideation and planning with 19 items scaled from 0 (least severe) to 2 (most severe), and a possible total score ranging from 0 to 38..
  units on a scale | 15.7 (6.9) | 14.3 (6.3) | 14.98 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Scale for Suicidal Ideation
Description: Change in suicidal ideation in depressed patients with moderate to severe suicidal thoughts from the pre-infusion baseline to 24 hours after the infusion with ketamine or midazolam, a sedative not known to reduce suicidal ideation, measured with Beck Scale for Suicidal Ideation - clinician rated version. This scale has 19 items scaled 0 (least severe) to 2 (most severe) and a potential score ranging from 0 to 38, with higher score indicating greater severity.
Time Frame: Day 1 (24 hours) post-treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Midazolam | Ketamine
Number analyzed (Participants) | 40 | 40
units on a scale | -3.66 (0.93) | -8.62 (0.93)

2. Secondary Outcome: Saliva Cortisol Awakening Response (CAR).
Description: On the mornings of an infusion day and on post-treatment day1, participants used salivettes (Sarstedt AG & Co.) to provide saliva samples upon awakening (Cort1) and 30 minutes later (Cort2) to measure cortisol awakening response (CAR) = (Cort2 - Cort1).
  Differences between the midazolam and ketamine groups were tested using an analysis of covariance (ANCOVA) model of the change in CAR from baseline to day1, with treatment group and baseline measurement of the outcome variable as predictors.
  Range from 0.1 to 12.5 ng/ml and lower means less stress response, higher means greater stress response.
Time Frame: Cort2 - Cort1 = (Day 1 30-mins post-awakening cortisol) - (Day 1 awakening cortisol)
Measure: Mean (Standard Deviation); unit: log(ng/mL)
Arm/Group | Midazolam | Ketamine
Number analyzed (Participants) | 40 | 40
log(ng/mL)
  Baseline awakening | 0.94 (0.61) | 0.47 (1.16)
  Baseline 30 mins post-awakening | 1.29 (0.53) | 0.88 (1.17)
  Day1 awakening | 0.77 (0.76) | 0.74 (0.88)
  Day1 30 minutes post-awakening | 1.19 (0.74) | 1.06 (0.84)

3. Secondary Outcome: Neuropsychological Effects
Description: The average Z-scores reported below are the average of the Z-scores for all tests administered. The Z-scores for each test were based on published normative data and normative data available in our laboratory. The population mean for a Z-score is zero, with a SD of 1, thus scores below zero would indicate performance below the population norm; a score close to zero indicates performance close to the population norm (or a normalizing of performance).
Time Frame: Baseline and Day 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Midazolam | Ketamine
Number analyzed (Participants) | 40 | 40
score on a scale
  Pre-infusion overall neuropsych performance | -0.252 (0.096) | -0.306 (0.096)
  Day1 post-infusion overall neuropsych performance | -0.146 (0.106) | -0.01 (0.106)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the 24 hour primary outcome study period.
Description: For the other (not including serious) adverse events, the total numbers without specific types, are reported here, with further detail available in the published paper.
Arm/Group | Midazolam | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 4/40 | 5/40
Other Adverse Events (participants affected / at risk) | 12/40 | 10/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=40) | Ketamine (N=40)
Inpatient admission for suicidal ideation (General disorders) | 2 (2) | 1 (1)
overdose (General disorders) | 2 (2) | 3 (3)
medical illness unrelated to study (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=40) | Ketamine (N=40)
Subjects with any event (General disorders) | 12 (13) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT01700829/Prot_000.pdf